CLINICAL TRIAL: NCT04365842
Title: Development, Feasibility, and Effectiveness of Smartphone Application for Hand Therapy for Patients With Rheumatoid Arthritis: Mix Method Study
Brief Title: Effectiveness of Technology-Supported Hand Strengthening and Stretching Exercises in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Eda Tonga, Assoc. Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 09.2019.577
Record Dates: First submitted 2020-04-15; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Rheumatoid Arthritis
Keywords: mhealth; hand exercise; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital exercise group (Experimental): After the 6-week digital intervention, 1) qualitative interviews have done with 6-15 patients from intervention group to assess the feasibility of digital intervention.
  2) The primary outcomes are hand pain and function and exercise adherence will be evaluated for all participants
  Interventions: Behavioral: Digital exercise group
- Waiting list conrol (Active Comparator): A hand rehabilitation home program will be given to the patients in the group through the telephone messages with brochures.
  Interventions: Other: General Home Hand Therapy

INTERVENTIONS:
Behavioral: Digital exercise group — Hand Rehabilitation Program: Developed hand exercise smartphone app which include: Self-assessment, (b) self-monitoring (c) exercises types/frequency/ diary, (d) patient education, (e) behavioral change and encouragement (f) exercise adherence Sample exercises
  1. Hand and finger movements: 6-8 repetitions, according to the diagnosis of the patient
  2. Strengthening exercises of hand and finger muscles
  3. Exercises to increase grip and pinch strength
  4. Exercises to increase tendon swing and pull angle
  Arms: Digital exercise group
Other: General Home Hand Therapy — Hand rehabilitation home program will be given to the through the telephone messages with brochures.
  1. Hand and finger movements: 6-8 repetitions, according to the diagnosis of the patient
  2. Strengthening exercises of hand and finger muscles
  3. Exercises to increase grip and pinch strength
  4. Exercises to increase tendon swing and pull angle
  Arms: Waiting list conrol

SUMMARY:
Growing research evidence supports the effectiveness of mHealth interventions for improving exercise adherence and motivation. The aims of our study are; 1) to develop and design a smartphone application for a structured hand exercise program for patients with RA and to test its usability. 2) Evaluate the feasibility and effectiveness of hand exercise app. This study is a mixed-methods study that aims to investigate the effectiveness of the Mar-HandTherapy app: a qualitative and quantitative study with the iterative design approach.

DETAILED DESCRIPTION:
The long-term beneficial effects of strengthening and stretching for rheumatoid arthritis (RA) for hand programs (SARAH) on functions have been shown in recent studies. Also, recently a usable web-based hand exercise program developed for patients with RA in UK. 1- The aim of our study is to develop and design a smartphone application for structured hand exercise program for patients with RA and to test its usability. 2- Evaluate the feasibility and effectiveness of smartphone app hand exercise app. In our study, a qualitative iterative design approach that includes focus groups of experts/patients was used. The mobile application was designed in 3 phases: PHASE 1: we conducted focus group meetings to compromise the content, feature and design of app in the first phase (Prototype version of smartphone software for RA hand training program/Mar-Hand-Therapy app). Focus Group were consisted two physiotherapist (PT), three hand therapists (HT) working in the field in different rheumatology or hand rehabilitation clinics, two software-computer engineers, 3 patients with RA who had previously participated hand therapy. All focus group members (n=10) and 6 patients used the app for one week. All users filled the usability questionnaire, made the comments and advises. The revised version was tested again for one week. The last revised version completed after two weeks tested. 40 patients diagnosed with rheumatoid arthritis will be included to the study. Participants randomized to digital intervention and waiting list control. After the 6-week digital intervention qualitative interviews have done with 6-15 patients from intervention group to assess the feasibility of digital intervention. The primary outcomes are hand pain and function and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with rheumatoid arthritis according to ARA criteria
* RA patients with stage 2 or 3 according to ACR criteria
* The first symptoms started at least a year ago and those who are undergoing medical treatment
* Those between the ages of 18-65

Exclusion Criteria:

* Those who are in the inflammatory period
* Those who have had surgery for neurological, orthopedic or other reasons recently
* Those with specified depression or other psychological diagnosis
* Those who have received physiotherapy and ergotherapy in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Hand pain at 7 week | Baseline and week 7
  Measurement of health perspective with 100 mm visual analogue scale (VAS). We assess the hand pain score change from baseline scores at 7th week.
  The leftmost value in the 100mm horizontal line used for VAS is scored between 0 mm (no pain) and the rightmost value is rated between 100mm (unbearable pain).
exercise adherance | week 7
  Qualitative data from smartphone (Time using the app, times of using videos etc)

SECONDARY OUTCOMES:
Change from baseline of Hand Function | Baseline and week 7
  Measure of Activity Performance in the Hand (MAP-HAND). It consists of 18 questions. Each question scores between 0 and 3 points. It worsens as the total score increases.We assess the hand function score change from baseline. scores at 7th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Argent R, Daly A, Caulfield B. Patient Involvement With Home-Based Exercise Programs: Can Connected Health Interventions Influence Adherence? JMIR Mhealth Uhealth. 2018 Mar 1;6(3):e47. doi: 10.2196/mhealth.8518. PMID 29496655
- [Background] Srikesavan CS, Williamson E, Eldridge L, Heine P, Adams J, Cranston T, Lamb SE. A Web-Based Training Resource for Therapists to Deliver an Evidence-Based Exercise Program for Rheumatoid Arthritis of the Hand (iSARAH): Design, Development, and Usability Testing. J Med Internet Res. 2017 Dec 13;19(12):e411. doi: 10.2196/jmir.8424. PMID 29237581
- [Background] Azevedo R, Bernardes M, Fonseca J, Lima A. Smartphone application for rheumatoid arthritis self-management: cross-sectional study revealed the usefulness, willingness to use and patients' needs. Rheumatol Int. 2015 Oct;35(10):1675-85. doi: 10.1007/s00296-015-3270-9. Epub 2015 Apr 24. PMID 25903352
- [Background] Choi W, Zheng H, Franklin P, Tulu B. mHealth technologies for osteoarthritis self-management and treatment: A systematic review. Health Informatics J. 2019 Sep;25(3):984-1003. doi: 10.1177/1460458217735676. Epub 2017 Nov 1. PMID 29090628